CLINICAL TRIAL: NCT03375008
Title: Development of Non-invasive Magnetic Resonance Imaging Diagnostic Method for Nonalcoholic Steatohepatitis(NASH)
Brief Title: Predictable MR Index for Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Chang Hee Lee, Professor, Korea University Guro Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KUGH16184
Record Dates: First submitted 2017-11-22; First posted 2017-12-15 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Magnetic resonance imager(MRI); Nonalcoholic fatty liver disease(NAFLD); Imaging diagnostic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diagnostic Imaging; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging diagnostic and biopsy (Experimental): 47 subjects who are suspected NASH from June 2016 to December 2017.
  Interventions: Diagnostic Test: Imaging diagnostic and biopsy

INTERVENTIONS:
Diagnostic Test: Imaging diagnostic and biopsy — Liver biopsy and MRI scan

SUMMARY:
1. To evaluate feasibility of using multiparametric Magnetic resonance(MR) imaging to predict nonalcoholic steatohepatitis(NASH)
2. To develop non-invasive diagnosis tool using multiparametric Magnetic resonance(MR) imaging for nonalcoholic steatohepatitis(NASH)

DETAILED DESCRIPTION:
Nonalcoholic steatohepatitis(NASH) is a severe form of nonalcoholic fatty liver disease(NAFLD). The causes are known to be associated with metabolic diseases such as obesity, insulin resistance type 2 diabetes, and hypercholesterolemia. Histologically, it is characterized by steatosis, hepatocellular injury, and inflammation and fibrosis of the liver parenchyma. Nonalcoholic steatohepatitis (NASH) may progress to cirrhosis and hepatocellular carcinoma(HCC) may develop even in patients without viral hepatitis, therefore there have been much interest and many researches in causation and diagnosis for nonalcoholic steatohepatitis(NASH).

Liver biopsy remains the gold standard for the diagnosis of nonalcoholic fatty liver disease(NAFLD) and is the only reliable method for differentiating nonalcoholic steatohepatitis(NASH) from simple steatosis. However, liver biopsy has several drawbacks, including invasiveness, potential complications such as excessive bleeding and death, sampling error, and inter- and intra-observer variability.

Magnetic resonance(MR) imaging has been used as a multiparametric imaging tool with which to evaluate steatosis by chemical shift imaging andm magnetic resonance(MR) spectroscopy, and fibrosis by magnetic resonance(MR) elastography and T1 mapping. To the best of our knowledge, there is no accurate imaging diagnostic tool for nonalcoholic steatohepatitis(NASH), therefore the investigators aimed to develop non-invasive imaging diagnostic model using multiparametric magnetic resonance imager(MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Patients >19 years age
2. Patients who had elevated aspartate transaminase(AST)/alanine transaminase(ALT) and fatty liver on abdominal ultrasonography
3. Patients who are clinically suspected to have nonalcoholic steatohepatitis(NASH)

   * Clinically suspected nonalcoholic steatohepatitis(NASH): >40 years age, metabolic syndrome, fibrosis on transient elastography(TE, Fibroscan), or elevated Fibrosis-4(FIB-4), Aspartate aminotransferase-to-platelet ratio index(APRI), nonalcoholic fatty liver disease fibrosis score(NFS) on blood tests
4. Patients who underwent (<6 months) or will undergo US-guided liver biopsy

Exclusion Criteria:

1. Chronic liver disease other than nonalcoholic fatty liver disease(NAFLD) (chronic hepatitis B or C, autoimmune hepatitis, primary biliary sclerosis)
2. Alcohol abuse (men, >140g/week; women, >70g/week)
3. Fatty liver due to medication
4. Contraindication to magnetic resonance imager(MRI)
5. Hepatocellular carcinoma
6. Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Radiologic Diagnosis & Criteria of nonalcoholic steatohepatitis(NASH) | up to 23 month
  Development of non-invasive magnetic resonance imaging diagnostic model for NASH using linear regression analysis
  1. Linear regression analysis using three magnetic resonance(MR) parameters 1) Fat signal fraction measured on MR spectroscopy (unit: %) 2) Liver stiffness measured on MR elastography (unit: kPa) 3) T1 relaxation time measured on T1 mapping (unit: msec) → Development of linear equation for NAFLD activity score (NAS) and Steatosis, Activity, Fibrosis (SAF) score
  2. Fitting of observed values (NAS, SAF score) and predicted values (NAS, SAF score) → Obtaining R square (R2) (Unit: none)

SECONDARY OUTCOMES:
Fat imaging : Fat signal fraction measured on magnetic resonance(MR) spectroscopy | During scanning, up to 15 seconds
  * Fat signal fraction measured on magnetic resonance(MR) spectroscopy
  1. high speed T2-corrected multi-echo (HISTO) MR spectroscopic technique
     * multiple short echo time : correction of T2 bias
     * long repetition time: correction of T1 bias
  2. 15 x 15 x 15-mm square-shaped region-of-interest(ROI) → Right hepatic lobe
  3. 3 times measurement → mean value was used as a representative value
  4. unit: percentage (%)
  5. Receiver operating characteristic (ROC) curve analysis for steatosis grade (0-3) → Obtaining cut-off values of each steatosis grade and area under the curve (AUC)
Fibrosis imaging(1) : Liver stiffness measured on magnetic resonance elastography(MRE) | During scanning, up to 20 seconds
  * Magnetic resonance elastography(MRE)
  1. 60 Hz acoustic wave
  2. Four slices were obtained for each magnetic resonance elastography(MRE) examination
  3. Stiffness maps (elastograms) for each magnetic resonance elastography(MRE) slices were automatically generated
  4. free-hand region-of-interest (ROI) on the right hepatic lobe
  5. 5 times measurement → mean value was used as a representative value
  6. unit: kilopascal (kPa)
  7. Receiver operating characteristic (ROC) curve analysis for fibrosis grade (0-4) → Obtaining cut-off values of each fibrosis grade and area under the curve (AUC)
Fibrosis imaging(2) : T1 relaxation time measured on T1 mapping | During scanning, up to 20 seconds
  * T1 mapping
  1. Shortened Modified Look Locker Inversion (shMOLLI) recovery sequence
  2. Four slices were obtained for each T1 map
  3. Oval-shaped region-of-interest (ROI) in the right hepatic lobe
  4. 5 times measurement → mean value was used as a representative value
  5. unit: millisecond (msec)
  6. Receiver operating characteristic (ROC) curve analysis for ballooning (0-2), lobular inflammation (0-3), fibrosis grade (0-4) → Obtaining cut-off values of each grade and area under the curve (AUC)
Histologic interpretation(1) : Nonalcoholic fatty liver disease activity score (NAS) | Up to a week
  1. the sum of each histological component semiquantitatively evaluated as follows: steatosis (0-3), ballooning (0-2), and lobular inflammation (0-3)
  2. NAS 0-2: not considered steatohepatitis
  3. NAS 3-4: possible steatohepatitis 4/ NAS ≥5: definite steatohepatitis
Histologic interpretation(1) : Steatosis, Activity, Fibrosis (SAF) score | Up to a week
  1. steatosis (0-3), ballooning degeneration (0-2), lobular inflammation (0-2), and fibrosis (0-4).
  2. Nonalcoholic steatohepatitis(NASH): when steatosis is present and when both features of activity (ballooning and lobular inflammation) display at least grade 1
  3. Unit: None

CONTACTS AND LOCATIONS:
Overall Officials: Chang Hee Lee, MD, Ph.D., Principal Investigator — Professor
Locations (1):
- Korea University Guro Hospital, Seoul, Guro-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-23. doi: 10.1002/hep.25762. No abstract available. PMID 22488764
- [Background] Poynard T, Lenaour G, Vaillant JC, Capron F, Munteanu M, Eyraud D, Ngo Y, M'Kada H, Ratziu V, Hannoun L, Charlotte F. Liver biopsy analysis has a low level of performance for diagnosis of intermediate stages of fibrosis. Clin Gastroenterol Hepatol. 2012 Jun;10(6):657-63.e7. doi: 10.1016/j.cgh.2012.01.023. Epub 2012 Feb 14. PMID 22343514
- [Background] Banerjee R, Pavlides M, Tunnicliffe EM, Piechnik SK, Sarania N, Philips R, Collier JD, Booth JC, Schneider JE, Wang LM, Delaney DW, Fleming KA, Robson MD, Barnes E, Neubauer S. Multiparametric magnetic resonance for the non-invasive diagnosis of liver disease. J Hepatol. 2014 Jan;60(1):69-77. doi: 10.1016/j.jhep.2013.09.002. Epub 2013 Sep 12. PMID 24036007
- [Background] Park YS, Lee CH, Kim JH, Kim BH, Kim JH, Kim KA, Park CM. Effect of Gd-EOB-DTPA on hepatic fat quantification using high-speed T2-corrected multi-echo acquisition in (1)H MR spectroscopy. Magn Reson Imaging. 2014 Sep;32(7):886-90. doi: 10.1016/j.mri.2014.04.010. Epub 2014 Apr 24. PMID 24853467
- [Background] Ishak K, Baptista A, Bianchi L, Callea F, De Groote J, Gudat F, Denk H, Desmet V, Korb G, MacSween RN, et al. Histological grading and staging of chronic hepatitis. J Hepatol. 1995 Jun;22(6):696-9. doi: 10.1016/0168-8278(95)80226-6. No abstract available. PMID 7560864
- [Background] Brunt EM, Janney CG, Di Bisceglie AM, Neuschwander-Tetri BA, Bacon BR. Nonalcoholic steatohepatitis: a proposal for grading and staging the histological lesions. Am J Gastroenterol. 1999 Sep;94(9):2467-74. doi: 10.1111/j.1572-0241.1999.01377.x. PMID 10484010
- [Background] SCHEUER PJ, WILLIAMS R, MUIR AR. Hepatic pathology in relatives of patients with haemochromatosis. J Pathol Bacteriol. 1962 Jul;84:53-64. No abstract available. PMID 14498313
- [Background] Kleiner DE, Brunt EM, Van Natta M, Behling C, Contos MJ, Cummings OW, Ferrell LD, Liu YC, Torbenson MS, Unalp-Arida A, Yeh M, McCullough AJ, Sanyal AJ; Nonalcoholic Steatohepatitis Clinical Research Network. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology. 2005 Jun;41(6):1313-21. doi: 10.1002/hep.20701. PMID 15915461
- [Background] Piechnik SK, Ferreira VM, Dall'Armellina E, Cochlin LE, Greiser A, Neubauer S, Robson MD. Shortened Modified Look-Locker Inversion recovery (ShMOLLI) for clinical myocardial T1-mapping at 1.5 and 3 T within a 9 heartbeat breathhold. J Cardiovasc Magn Reson. 2010 Nov 19;12(1):69. doi: 10.1186/1532-429X-12-69. PMID 21092095